CLINICAL TRIAL: NCT05830149
Title: A Prospective Randomized, Controlled Clinical Trial on the Efficacy of Cryoinsufflation for the Treatment of Hidradenitis Suppurativa
Brief Title: Safety and Treatment of Cryoinsufflation in Treatment of Hidradenitis Suppurativa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not have staffing to support the study
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB11587
Record Dates: First submitted 2022-01-27; First posted 2023-04-26 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either receiving cryoinsufflation or surgical deroofing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoinsufflation (Experimental): In cryoinsufflation, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar local anesthetic. A needle will be mounted on a liquid nitrogen cryosurgical unit. The needle will be inserted through the entire sinus tract and cryospray will be delivered to the length of the sinus tract as the needle is retracted with the intention to induce local tissue destruction. Each spray will be 5 seconds in duration and each tract will be sprayed 3 times per treatment session. This technique has been shown to be effective in sinus tract obliteration. This intervention may prevent local disease progression and prevent patients from undergoing more invasive surgeries. Overall, this would result in improved cosmesis, decreased pain, decreased bleeding and improved patient satisfaction.
  Interventions: Other: Cryoinsufflation
- Deroofing (Active Comparator): Deroofing will serve as the control group as this is a minimally invasive procedure that is used for sinus tracts in HS. Studies have demonstrataed the efficacy of deroofing in treating the draining sinus tracts in HS. The control group should have decreased drainage, pain, recurrence, and scarring. In deroofing, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar local anesthetic. The sinus tract is probed to clearly defined the sinus tract. The skin overlying the sinus tract is cut using an a scalpel. In this way, the top of the sinus tract is surgically removed. In this way, the top of the sinus tract is surgically removed. The floor of the sinus tract is exposed and left open to heal by secondary intention.
  Interventions: Other: Deroofing

INTERVENTIONS:
Other: Cryoinsufflation — In cryoinsufflation, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar local anesthetic. A needle will be mounted on a liquid nitrogen cryosurgical unit. The needle will be inserted through the entire sinus tract and cryospray will be delivered to the length of the sinus tract as the needle is retracted with the intention to induce local tissue destruction. Each spray will be 5 seconds in duration and each tract will be sprayed 3 times per treatment session. This technique has been shown to be effective in sinus tract obliteration. This intervention may prevent local disease progression and prevent patients from undergoing more invasive surgeries. Overall, this would result in improved cosmesis, decreased pain, decreased bleeding and improved patient satisfaction.
  Arms: Cryoinsufflation
Other: Deroofing — Deroofing will serve as the control group as this is a minimally invasive procedure that is used for sinus tracts in HS. Studies have demonstrataed the efficacy of deroofing in treating the draining sinus tracts in HS. The control group should have decreased drainage, pain, recurrence, and scarring. In deroofing, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar local anesthetic. The sinus tract is probed to clearly defined the sinus tract. The skin overlying the sinus tract is cut using an a scalpel. In this way, the top of the sinus tract is surgically removed. In this way, the top of the sinus tract is surgically removed. The floor of the sinus tract is exposed and left open to heal by secondary intention.
  Arms: Deroofing

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic, socially and cosmetically debilitating disease. It typically manifests as nodules and abscesses that ultimately can progress to form deep sinus tracts, fistulas, and scarring. The lesions are often very painful and can chronically drain malodorous fluid, which can leave affected individuals uncomfortable and self-conscious, or even debilitated. Treatment presents significant challenges and frustration to both the patient and the provider. Measures such as topical antibiotic and antiseptic washes are generally thought to be beneficial for the treatment of early stage HS. When this is not efficacious, systemic antibiotics are prescribed. In some patients, disease remains refractory to these treatments and their fistulas and tracts progress to scarring. In some patients, the disease continues to progress. In these patients who fail conservative medical management and minimally invasive procedures, such as deroofing, is the next step in the therapeutic ladder. In deroofing, the skin overlying the sinus tract is cut, exposing the floor of the tract. These wounds are left open to heal by secondary intention. Also with this technique, recurrence is common.

In this study, investigators propose the use of cryoinsufflation for management of the sinus tracts in hidradenitis suppurativa. In this technique, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar numbing medication. A needle will be mounted on a cryosurgical unit. The needle will be instered into the tracts at one location on one side of the body and liquid nitrogen will be administered. This will result in obliteration of the sinus tract. This intervention may prevent disease progression and ameliorate the need for these patients to surgically intervene on their disease. Overall, this would result in improved cosmesis, decreased pain, and improved patient satisfaction. The objective of this prospective, randomized controlled clinical trial is to compare the efficacy of cryoinsufflation in patients with draining sinus tracts versus deroofing while keeping the patients on the medications that they currently on for hidradenitis suppurativa.

In deroofing, the sinus tract is found. Local anesthesia is administered to numb the area of the sinus tract. The sinus tract is probed. Then the skin overlying the sinus tract is cut, exposing the floor of the tract. These wounds are then left open to heal by secondary intention.

Patients with one anatomic location having Hurley stage 2 disease with at least one recurrent sinus tract will be included in the study. Cryoinsufflation will be compared to deroofing. Patients will be randomized into either the group receiving cryoinsufflation (Group A) or deroofing (Group B). The distribution of patients will be completely random similar to a coin toss. Patients will remain on all systemic hidradenitis suppurativa medications throughout the entire duration of the study. The primary endpoint of the study will be time to obliteration of the sinus tract and pain tolerance of cryoinsufflation. Secondary endpoints will include cosmesis (identified through patient photography) and patient satisfaction (identified through study surveys) as well as comparison to deroofing. Patients in group A will be treated with cryoinsufflation at up to five study visits. If it is determined that the patient's sinus tract has scarred over, that will be the patient's final study visit and cryoinsufflation will not be performed. Patients in group B will be treated with deroofing at the first visit and will return for 2 future visits at 28 day intervals. At the study visits the investigators will examine the site of intervention, take clinical photographs, measure the tract, ultrasound the tract, the study doctor will perform visual assesments of the area, the interventions (both cryoinsufflation and deroofing) will be timed, and patients will complete the survey questionnaires. If determined to be superior in efficacy, the addition of cryoinsufflation as an adjuvant therapy to hidradenitis suppurativa could influence treatment guidelines in hidradenitis management, leading to an improvement in the quality of care delivered, especially in terms of cosmetic outcomes, prevention of disease progression, and patient satisfaction.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, socially and cosmetically debilitating disease. It typically manifests as nodules and abscesses that ultimately can progress to form deep sinus tracts, fistulas, and scarring. The lesions are often very painful and can chronically drain malodorous fluid, which can leave affected individuals uncomfortable and self-conscious, or even debilitated. Treatment presents significant challenges and frustration to both the patient and the provider. Measures such as topical antibiotic and antiseptic washes are generally thought to be beneficial for the treatment of early stage HS. When this is not efficacious, systemic antibiotics are prescribed. In some patients, disease remains refractory to these treatments and their fistulas and tracts progress to scarring. In some patients, the disease continues to progress. In these patients who fail conservative medical management and minimally invasive procedures, such as deroofing, is the next step in the therapeutic ladder. The edge of the incised wounds quickly achieved epithelialization through secondary intention healing. In deroofing, the skin overlying the sinus tract is cut, exposing the floor of the tract. These wounds are left open to heal by secondary intention. Also in this technique, recurrence is common.

The Hurley Staging system is commonly utilized to classify the severity of a patient's hidradenitis suppurativa. Stage 1 disease consists of one or more abscesses with no sinus tract formation or scarring. Stage 2 disease involves one or more widely separated recurrent abscesses, with formation of a sinus tract and/or scarring. Stage 3 involves multiple interconnected sinus tracts and/or abscesses throughout an anatomical area.

In this study, investigators propose the use of cryoinsufflation for management of the sinus tracts in Hurley stage 2 hidradenitis suppurativa as a faster, less invasive means of treating HS compared to deroofing. In this technique, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar local anesthetic. A needle will be mounted on a liquid nitrogen cryosurgical unit. The needle will be inserted through the entire sinus tract and cryospray will be delivered to the length of the sinus tract as the needle is retracted with the intention to induce local tissue destruction. Each spray will be 5 seconds in duration and each tract will be sprayed 3 times per treatment session. This technique has been shown to be effective in sinus tract obliteration. This intervention may prevent local disease progression and prevent patients from undergoing more invasive surgeries. Overall, this would result in improved cosmesis, decreased pain, decreased bleeding and improved patient satisfaction. The objective of this prospective, randomized controlled clinical trial is to compare the efficacy of cryoinsufflation in patients with draining sinus tracts versus the treatment that the patient is currently on for hidradenitis suppurativa.

Deroofing will serve as the control group as this is a minimally invasive procedure that is used for sinus tracts in HS. Studies have demonstrataed the efficacy of deroofing in treating the draining sinus tracts in HS. The control group should have decreased drainage, pain, recurrence, and scarring. In deroofing, local anesthesia will be administered to the tract area with lidocaine hydrochloride 1% or a similar local anesthetic. The sinus tract is probed to clearly defined the sinus tract. The skin overlying the sinus tract is cut using an a scalpel. In this way, the top of the sinus tract is surgically removed. In this way, the top of the sinus tract is surgically removed. The floor of the sinus tract is exposed and left open to heal by secondary intention.

Patients with hidradenitis suppurativa with at least one anatomic location having Hurley stage 2 hidradenitis suppurativa will be included in the study. Cryoinsufflation will be compared to deroofing, currently a widely used modality for sinus tract destruction. Patients will be randomized into either the group receiving cryoinsufflation or deroofing. The distribution of patients will be completely random similar to a coin toss. The investigators will write "group A" on 10 pieces of paper and "group B" on 10 pieces of paper. When enrolling a new patient, investigators will draw one slip of paper. If the slip of paper says "group A" the patient will be in the cryoinsufflation arm of the study. If the slip of paper says "group B", the patient will be in the deroofing arm of the study. Patients will remain on all systemic hidradenitis suppurativa medications throughout the entire duration of the study.

The primary endpoint of the study will be time to obliteration of the sinus tract and pain of cryoinsufflation. Secondary endpoints will include cosmesis (identified through patient photography) and patient satisfaction (identified through study surveys). Patients in Group A will be treated with cryoinsufflation at up to 5 study visits and will return for one post-treatment study visit 28 days after the last treatment with cryoinsufflation. Patients in Group B will be treated with deroofing at 1 study visit and will return for two post-treatment study visits at 28 day intervals. At the study visits the investigators will examine the site of intervention, take clinical photographs, measure the tract, ultrasound the tract, the study doctor will perform visual assesments of the area, the interventions (both cryoinsufflation and deroofing) will be timed, and patients will complete the survey questionnaires. If determined to be superior in efficacy, the addition of cryoinsufflation as an adjuvant therapy to hidradenitis suppurativa could influence treatment guidelines in hidradenitis suppurativa management, leading to an improvement in the quality of care delivered, especially in terms of cosmetic outcomes, prevention of disease progression, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old.
2. Have a diagnosis of HS.
3. Patients must HS with one anatomic location being Hurley stage 2 disease, with one or more widely separated, recurrent sinus tracts.
4. Sinus tracts must measure < 5 cm in length.
5. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form.
6. Agree to follow and undergo all study-related procedures.

Exclusion Criteria:

1. Patients who are pregnant or breast feeding will not be able to take part in the study due to the unknown effects of cryoinsufflation.
2. Any reason the investigator feels the patient should not participate in the study.
3. If a patient misses ≥ 2 consecutive study visits, the patient will be excluded from further participation in this trial.
4. Patients who have a history of keloid scarring.
5. Patients planning to undergo surgery intervention for hidradenitis suppurativa during the study period.
6. Patients with a history of kidney or liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Vancouver scar scale to assess efficacy of 1 treatment session every 28 days for up to 5 treatments | At the end of Cycle 1 (each cycle is 28 days)
  Scars will be assessed using The Vancouver Scar Scale. Pigmentation, vascularity, pliability and height will be assessed and assigned a rating using the following:
  Pigmentation (0-2) Normal (0) Hypopigmentation (1) Hyperpigmentation (2)
  Vascularity (0-3) Normal (0) Pink (1) Red (2) Purple (3)
  Pliability (0-5) Normal (0) Supple (1) Yielding (2) Firm (3) Banding (4) Contracture (5)
  Height (0-3) Normal (flat) (0) 0-2 mm (1) 2-5 mm (2) >5 mm (3)

SECONDARY OUTCOMES:
Quality of life changes secondary to study intervention with the DLQI (Dermatology Quality of Life Index) questionnaire | At the end of Cycle 1 (each cycle is 28 days)
  2. To determine any changes in quality of life in patients participants every 28 days
  DLQI Scoring
  SCORING
  The scoring of each question is as follows:
  Very much, scored 3 A lot scored, 2 A little scored, 1 Not at all scored, 0 Not relevant scored, 0 Question 7, 'prevented work or studying', scored 3
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
  DLQI SCORE INTERPRETATION 0 - 1 no effect at all on patient's life 2 - 5 small effect on patient's life 6 - 10 moderate effect on patient's life 11 - 20 very large effect on patient's life 21 - 30 extremely large effect on patient's life
Safety - adverse event assessment | At the end of Cycle 1 (each cycle is 28 days)
  3. Participants will be evaluated at each visit to assess for adverse events.
Hurley Staging assessment | At the end of Cycle 1 (each cycle is 28 days)
  Participant treatment location will be assessed using the Hurley Staging scale
  Stage I (Mild) Inflammatory nodule or abscess formation, single or multiple, without sinus tracts and scarring
  Stage II (Moderate) Recurrent abscesses and nodules with sinus tract formation or scarring: single or multiple widely separated lesions
  Stage III (Severe) Diffuse or near-diffuse involvement with multiple interconnected sinus tracts, scarring, and abscesses across entire area

CONTACTS AND LOCATIONS:
Overall Officials: Pranita Rambhatla, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No